CLINICAL TRIAL: NCT02595879
Title: Phase I Dose-Escalation Bioavailability Study of Oral Triapine in Combination With Concurrent Chemoradiation for Locally Advanced Cervical Cancer (LACC) and Vaginal Cancer
Brief Title: Triapine With Chemotherapy and Radiation Therapy in Treating Patients With IB2-IVA Cervical or Vaginal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01907; NCI-2015-01907 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCC 15-157; UPCI 15-157; 15-157; 9892 (Other: UPMC Hillman Cancer Center LAO); 9892 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2024-10-16 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cervical Adenocarcinoma; Advanced Cervical Adenosquamous Carcinoma; Advanced Cervical Squamous Cell Carcinoma; Advanced Vaginal Adenocarcinoma; Advanced Vaginal Adenosquamous Carcinoma; Advanced Vaginal Squamous Cell Carcinoma; Stage IB2 Cervical Cancer AJCC v6 and v7; Stage II Cervical Cancer AJCC v7; Stage II Vaginal Cancer AJCC v6 and v7; Stage III Vaginal Cancer AJCC v6 and v7; Stage IIIB Cervical Cancer AJCC v6 and v7; Stage IVA Cervical Cancer AJCC v6 and v7; Stage IVA Vaginal Cancer AJCC v6 and v7
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Specimen Handling; Brachytherapy; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Congresses as Topic; Radiation; Fluorodeoxyglucose F18; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (triapine, chemoradiation) (Experimental): Patients undergo pelvic EBRT or IMRT 5 days per week for 5 weeks (25 fractions) with a 3-day boost in week 6, and 1 or 2 applications of LDR brachytherapy in week 6 or 5 fractions of HDR brachytherapy at week 4 or 5. Patients also receive triapine IV over 120 minutes on day 1 and PO on days 2-5, 8-12, 15-19, 22-26, and 29-33 within 90 minutes after pelvic irradiation, and cisplatin IV over 60-120 minutes once weekly for 5 weeks (days 2, 9, 16, 23, and 30). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients may receive a 6th cycle of cisplatin IV during the parametrial boost or any make-up radiation treatment in a sixth week of external beam radiotherapy. Patients undergo the collection of blood samples on study and undergo MRI and FDG-PET/CT during follow-up.
  Interventions: Procedure: Biospecimen Collection; Radiation: Brachytherapy; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Other: Fludeoxyglucose F-18; Radiation: High-Dose Rate Brachytherapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Other: Pharmacological Study; Procedure: Positron Emission Tomography; Drug: Triapine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Radiation: Brachytherapy — Undergo LDR brachytherapy
  Other Names: Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Internal Radiation Therapy; Radiation Brachytherapy; Radiation, Internal
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo FDG-PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: External Beam Radiation Therapy — Undergo pelvic EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Other: Fludeoxyglucose F-18 — Undergo FDG-PET/CT
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Radiation: High-Dose Rate Brachytherapy — Undergo HDR brachytherapy
  Other Names: Brachytherapy, High Dose; HDR; High dose brachytherapy (procedure)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Pharmacological Study — Correlative studies
Procedure: Positron Emission Tomography — Undergo FDG-PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Triapine — Given IV and PO
  Other Names: 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; 3-AP; 3-Apct; OCX-0191; OCX-191; OCX191; PAN-811

SUMMARY:
This phase I trial studies the side effects and best dose of triapine when given with radiation therapy and cisplatin in treating patients with stage IB2-IVA cervical or vaginal cancer. Triapine may stop the growth of cancer cells by blocking an enzyme needed for cell growth. Cisplatin is a drug used in chemotherapy that kills cancer cells by damaging their deoxyribonucleic acid (DNA) and stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Adding triapine to standard treatment with cisplatin and radiation therapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerable dose (MTD) and recommended phase II dose (RP2D) of oral triapine when used in combination with cisplatin plus radiation therapy.

II. To determine the oral bioavailability of triapine. III. To describe the pharmacokinetics (PK) of oral and intravenous triapine.

SECONDARY OBJECTIVES:

I. To determine whether the metabolic complete response (mCR) rate of oral triapine in combination with cisplatin chemoradiation using fludeoxyglucose F 18 (18F-FDG)-positron emission tomography (PET)/computed tomography (CT) at post-therapy (3-month) is at least 70%.

II. To determine clinical overall response rate, progression-free survival, and overall survival.

III. To determine the correlation of methemoglobin proportion (%) and triapine pharmacokinetic exposure.

EXPLORATORY OBJECTIVE:

I. To determine whether active human immunodeficiency virus (HIV) antiretroviral therapy impacts the antitumor activity of triapine.

OUTLINE: This is a dose-escalation study of triapine.

Patients undergo pelvic external beam radiation therapy (EBRT) or intensity modulated radiation therapy (IMRT) 5 days per week for 5 weeks (25 fractions) with a 3-day boost in week 6, and 1 or 2 applications of low dose rate (LDR) brachytherapy in week 6 or 5 fractions of high dose rate (HDR) brachytherapy at week 4 or 5. Patients also receive triapine intravenously (IV) over 120 minutes on day 1 and orally (PO) on days 2-5, 8-12, 15-19, 22-26, and 29-33 within 90 minutes after pelvic irradiation, and cisplatin IV over 60-120 minutes once weekly for 5 weeks (days 2, 9, 16, 23, and 30). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients may receive a 6th cycle of cisplatin IV during the parametrial boost or any make-up radiation treatment in a sixth week of external beam radiotherapy. Patients undergo the collection of blood samples on study and undergo magnetic resonance imaging (MRI) and FDG-PET/CT during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a new, untreated histologic diagnosis of stage IB2 (> 5 cm), II, IIIB, IIIC or IVA squamous, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix or stage II-IVA squamous, adenocarcinoma, or adenosquamous carcinoma of the vagina not amenable to curative surgical resection alone; the presence or absence of lymph node metastasis will be based on pre-therapy 18F-FDG PET/CT; the patient must be able to tolerate imaging requirements of an 18F-FDG PET/CT scan
* Age >= 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Life expectancy greater than 6 months
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hgb) >= 10.0 g/dL (blood transfusions to reach this amount are allowed)
* Serum creatinine =< 1.5 mg/dL to receive weekly cisplatin

  * If serum creatinine is between 1.5 and 1.9 mg/dL, patients are eligible for cisplatin if the estimated creatinine clearance (CCr) is > 30 ml/min (for the purpose of estimating the CCr, the formula of Cockcroft and Gault for females should be used)
* Total serum bilirubin =< 1.5 x upper limit of normal (ULN) (in patients with known Gilbert syndrome, a total bilirubin =< 3.0 x ULN, with direct bilirubin =< 1.5 x ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Able to take oral medication
* Not pregnant and not breastfeeding; the effects of triapine on the developing human fetus are unknown; for this reason as well as because heterocyclic carboxaldehydethiosemicarbazones and radiation are known to be teratogenic, women of child-bearing potential and men must agree to use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; patient must have documented negative urine pregnancy test must be resulted within 7 days before initiating protocol therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with triapine, breastfeeding should be discontinued if the mother is treated with triapine; these potential risks may also apply to other agents used in this study
* For HIV and hepatitis B/C (HEPB/C):

  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for the dose escalation portion of this trial; for those patients who are enrolled in the HIV positive (+) expansion cohort, they must be HIV infected and be on retroviral therapy with an undetectable viral load within 6 months of enrollment
  * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured; for patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Able to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patient has had a prior invasive malignancy diagnosed within the last three years (except [1] non-melanoma skin cancer or [2] prior in situ carcinoma of the cervix)
* Patients are excluded if they have received prior pelvic radiotherapy for any reason that would contribute radiation dose that would exceed tolerance of normal tissues at the discretion of the treating physician
* Patients receiving any other investigational agents
* Patients with known glucose-6-phosphate dehydrogenase deficiency (G6PD) are excluded due to an inability to administer the antidote for methemoglobinemia, methylene blue; pre-registration testing for G6PD is at the investigator's discretion and is not required for study enrollment
* Patients who are taking any medication associated with methemoglobinemia; medication must be discontinued and must have a washout period of 4 halflives or 4 weeks, whichever is shorter
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to triapine or cisplatin
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; known inadequately controlled hypertension; significant pulmonary disease including dyspnea at rest, patients requiring supplemental oxygen, or poor pulmonary reserve; or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with uncontrolled diabetes mellitus (fasting blood glucose controlled by medication, =< 200 mg/dL allowed)
* Patients who have had a hysterectomy or are planning to have an adjuvant hysterectomy following radiation as part of their cervical cancer treatment are ineligible
* Patients scheduled to be treated with adjuvant consolidation chemotherapy at the conclusion of their standard chemoradiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2026-04-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Taylor, Principal Investigator — University of Pittsburgh Cancer Institute LAO
Locations (17):
- United States (17):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor SE, Behr S, Cooper KL, Mahdi H, Fabian D, Gallion H, Ueland F, Vargo J, Orr B, Girda E, Courtney-Brooks M, Olawaiye AB, Randall LM, Richardson DL, Sullivan SA, Huang M, Christner SM, Beriwal S, Lin Y, Chauhan A, Chu E, Kohn EC, Kunos C, Ivy SP, Beumer JH. Dose finding, bioavailability, and PK-PD of oral triapine with concurrent chemoradiation for locally advanced cervical cancer and vaginal cancer (ETCTN 9892). Cancer Chemother Pharmacol. 2024 Dec 14;95(1):4. doi: 10.1007/s00280-024-04720-1. PMID 39673591

RESULTS

PARTICIPANT FLOW:
Groups:
- 100 mg PO Triapine + Chemoradiation; 150 mg PO Triapine + Chemoradiation: Patients undergo pelvic EBRT or IMRT 5 days per week for 5 weeks (25 fractions) with a 3-day boost in week 6, and 1 or 2 applications of LDR brachytherapy in week 6 or 5 fractions of HDR brachytherapy at week 4 or 5. Patients also receive triapine IV over 120 minutes on day 1 and 100mg PO on days 2-5, 8-12, 15-19, 22-26, and 29-33 within 90 minutes after pelvic irradiation, and cisplatin IV over 60-120 minutes once weekly for 5 weeks (days 2, 9, 16, 23, and 30). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients may receive a 6th cycle of cisplatin IV during the parametrial boost or any make-up radiation treatment in a sixth week of external beam radiotherapy. Patients undergo the collection of blood samples on study and undergo MRI and FDG-PET/CT during follow-up.
  Biospecimen Collection: Undergo collection of blood samples
  Brachytherapy: Undergo LDR brachytherapy
  Cisplatin: Given IV
  Computed Tomography: Undergo FDG-PET/CT
  External Beam Radiation Therapy: Undergo pelvic EBRT
  Fludeoxyglucose F-18: Undergo FDG-PET/CT
  High-Dose Rate Brachytherapy: Undergo HDR brachytherapy
  Intensity-Modulated Radiation Therapy: Undergo IMRT
  Magnetic Resonance Imaging: Undergo MRI
  Pharmacological Study: Correlative studies
  Positron Emission Tomography: Undergo FDG-PET/CT
  Triapine: Given IV and PO
Period: Cohort 1 / Dose Level 1
Arm/Group | 100 mg PO Triapine + Chemoradiation | 150 mg PO Triapine + Chemoradiation
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Cohort 2 / Dose Level 2
Arm/Group | 100 mg PO Triapine + Chemoradiation | 150 mg PO Triapine + Chemoradiation
Started | 0 | 4
Completed | 0 | 4
Not Completed | 0 | 0
Period: Cohort 3 / Dose Level 1
Arm/Group | 100 mg PO Triapine + Chemoradiation | 150 mg PO Triapine + Chemoradiation
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Expansion Cohort
Arm/Group | 100 mg PO Triapine + Chemoradiation | 150 mg PO Triapine + Chemoradiation
Started | 11 | 0
Completed | 10 | 0
Not Completed | 1 | 0
Not completed — Did not complete treatment regimen | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Triapine (100mg) + Chemoradiation): Patients undergo pelvic EBRT or IMRT 5 days per week for 5 weeks (25 fractions) with a 3-day boost in week 6, and 1 or 2 applications of LDR brachytherapy in week 6 or 5 fractions of HDR brachytherapy at week 4 or 5. Patients also receive triapine IV over 120 minutes on day 1 and PO on days 2-5, 8-12, 15-19, 22-26, and 29-33 within 90 minutes after pelvic irradiation, and cisplatin IV over 60-120 minutes once weekly for 5 weeks (days 2, 9, 16, 23, and 30). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients may receive a 6th cycle of cisplatin IV during the parametrial boost or any make-up radiation treatment in a sixth week of external beam radiotherapy. Patients undergo the collection of blood samples on study and undergo MRI and FDG-PET/CT during follow-up.
  Biospecimen Collection: Undergo collection of blood samples
  Brachytherapy: Undergo LDR brachytherapy
  Cisplatin: Given IV
  Computed Tomography: Undergo FDG-PET/CT
  External Beam Radiation Therapy: Undergo pelvic EBRT
  Fludeoxyglucose F-18: Undergo FDG-PET/CT
  High-Dose Rate Brachytherapy: Undergo HDR brachytherapy
  Intensity-Modulated Radiation Therapy: Undergo IMRT
  Magnetic Resonance Imaging: Undergo MRI
  Pharmacological Study: Correlative studies
  Positron Emission Tomography: Undergo FDG-PET/CT
  Triapine: Given IV and PO
- Triapine (150mg) + Chemoradiation): Patients undergo pelvic EBRT or IMRT 5 days per week for 5 weeks (25 fractions) with a 3-day boost in week 6, and 1 or 2 applications of LDR brachytherapy in week 6 or 5 fractions of HDR brachytherapy at week 4 or 5. Patients also receive triapine IV over 120 minutes on day 1 and PO on days 2-5, 8-12, 15-19, 22-26, and 29-33 within 90 minutes after pelvic irradiation, and cisplatin IV over 60-120 minutes once weekly for 5 weeks (days 2, 9, 16, 23, and 30). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients may receive a 6th cycle of cisplatin IV during the parametrial boost or any make-up radiation treatment in a sixth week of external beam radiotherapy. Patients undergo the collection of blood samples on study and undergo MRI and FDG-PET/CT during follow-up.
- Total: Total of all reporting groups
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation) | Total
Number analyzed (Participants) | 17 | 4 | 21
Age, Continuous [Median (Full Range); unit: years] | 51.0 [23.0 to 71.0] | 46.5 [35.0 to 56.0] | 51.0 [23.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 4 | 19
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 4 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Smoking History [Count of Participants; unit: Participants] — Smoking status at time of beginning study treatment = Yes / No / Unknown
  Participants
    Yes | 5 | 1 | 6
    No | 12 | 2 | 14
    Unknown | 0 | 1 | 1
Primary Site [Count of Participants; unit: Participants] — Original site of disease upon diagnosis
  Participants
    Cervix | 15 | 4 | 19
    Vagina | 2 | 0 | 2
Histology [Count of Participants; unit: Participants] — structures of cells and tissues classifications
  Participants
    adenocarcinoma | 3 | 2 | 5
    squamous cell carcinoma | 13 | 2 | 15
    adenosquamous | 1 | 0 | 1
Stage at Diagnosis [Count of Participants; unit: Participants] — IB: >5 mm limited to cervix II: beyond uterus, not extended to lower third of vagina or pelvic wall IIA: upper two-thirds of vagina no parametrial involvement IIB: Parametrial involvement not up to pelvic wall III: lower third of vagina and/or extends to pelvic wall and/or causes hydronephrosis or nonfunctioning kidney and/or involves pelvic and/or para-aortic lymph nodes; IIIB: Extends to pelvic wall and/or hydronephrosis or nonfunctioning kidney (unless due to other cause) IIIC: pelvic/para-aortic lymph nodes, despite tumor size/extent; lVA: adjacent pelvic organs IVB: distant organs
  Participants
    Stage IB | 1 | 1 | 2
    Stage II | 1 | 1 | 2
    Stage IIA | 1 | 0 | 1
    Stage IIB | 3 | 0 | 3
    Stage III | 1 | 1 | 2
    Stage IIIB | 1 | 0 | 1
    Stage IIIC | 7 | 1 | 8
    Stage IVA | 2 | 0 | 2
Stage [Count of Participants; unit: Participants] — I: Carcinoma strictly confined to the cervix 2: Invades beyond the uterus, but has not extended onto the lower third of the vagina or to the pelvic wall 3: Involves lower third of vagina and/or extends to the pelvic wall and/or causes hydronephrosis or nonfunctioning kidney and/or involves pelvic and/or para-aortic lymph nodes 4: Extends beyond the true pelvis or involves the mucosa of the bladder or rectum
  Participants
    Stage l | 1 | 1 | 2
    Stage ll | 5 | 1 | 6
    Stage lll | 9 | 2 | 11
    Stage lV | 2 | 0 | 2
ECOG [Count of Participants; unit: Participants] — ECOG PERFORMANCE STATUS
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    ECOG = 0 | 12 | 3 | 15
    ECOG = 1 | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was determined following a standard 3+3 design is as follows: Escalation at 0/3 DLTs, dose-reduction if >1/3 DLT, and expansion to 6 if 1/3 DLTs. DLT is defined as the severe toxicity event that leads to the termination of the treatment as defined in section 5.5. The highest dose level where <2/6 DLTs are observed will be declared MTD
Time Frame: Up to 5 weeks
Population: All treated patients evaluable for DLTs
Measure: Number; unit: mg
Groups:
- All Participants: Patients who received at least 80% of PO triapine (either at 100mg or 150mg) and 80% of chemoradiation.
Arm/Group | All Participants
Number analyzed (Participants) | 9
mg | 100

2. Primary Outcome: Number of Patients Who Experienced a DLT
Description: Number of patients that experienced a DLT, evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. DLTs are defined as the following adverse events if considered at least "possibly related" to a component of the study therapy and which occur from the start of treatment until completion of EBRT, prior to initiation of brachytherapy (i.e. the first 5 weeks if no treatments are missed): Any nausea, vomiting, diarrhea and elevation of serum creatinine level Grade 3 toxicity not resolved with maximal intervention to Grade 0-2 over 7 days (except alopecia and fatigue); Any nausea, vomiting, diarrhea and elevation of serum creatinine level Grade 4 toxicity; Any other non-hematologic toxicity ≥Grade 3; Any hematologic toxicity of ≥ Grade 4; Grade ≥3 dyspnea; Inability to deliver at least 20 of the scheduled 25 administrations of triapine at the planned dose, allowing for 2 weeks to make up missed radiation days.
  Inability to deliver
Time Frame: Up to 5 weeks
Population: All treated patients evaluable for DLTs
Measure: Count of Participants; unit: Participants
Groups:
- Triapine (100mg) + Chemoradiation): Patients undergo pelvic EBRT or IMRT 5 days per week for 5 weeks (25 fractions) with a 3-day boost in week 6, and 1 or 2 applications of LDR brachytherapy in week 6 or 5 fractions of HDR brachytherapy at week 4 or 5. Patients also receive triapine IV over 120 minutes on day 1 and 100mg PO on days 2-5, 8-12, 15-19, 22-26, and 29-33 within 90 minutes after pelvic irradiation, and cisplatin IV over 60-120 minutes once weekly for 5 weeks (days 2, 9, 16, 23, and 30).
- Triapine (150mg) + Chemoradiation): Patients undergo pelvic EBRT or IMRT 5 days per week for 5 weeks (25 fractions) with a 3-day boost in week 6, and 1 or 2 applications of LDR brachytherapy in week 6 or 5 fractions of HDR brachytherapy at week 4 or 5. Patients also receive triapine IV over 120 minutes on day 1 and 150mg PO on days 2-5, 8-12, 15-19, 22-26, and 29-33 within 90 minutes after pelvic irradiation, and cisplatin IV over 60-120 minutes once weekly for 5 weeks (days 2, 9, 16, 23, and 30).
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 6 | 3
Participants | 1 | 2

3. Primary Outcome: Bioavailability of Triapine
Description: The oral bioavailability of the oral form of the triapine will be measured as a numeric value using mass spectrophotometry.
Time Frame: Up to 2 weeks
Population: Patients that had both PO and IV triapine PK samples
Measure: Geometric Mean (95% Confidence Interval); unit: percentage
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 16 | 4
percentage | 60 [16 to 229] | 54 [15 to 200]

4. Primary Outcome: Cmax
Description: Maximum concentration
Time Frame: Up to 24 hours after dosing
Population: Treated patients for whom PK samples were able to be collected
Measure: Geometric Mean (Standard Deviation); unit: ug/L
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 17 | 4
ug/L | 476 (1.90) | 344 (1.91)

5. Primary Outcome: Tmax
Description: Time to maximum concentration,
Time Frame: Up to 24 hours after dosing
Population: Treated patients for whom samples were able to be collected
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 17 | 4
hours | 0.9 (3.0) | 1.5 (1.5)

6. Primary Outcome: AUC
Description: Area Under the Concentration-Time Curve (AUC 0-last)
Time Frame: Up to 24 hours after dosing
Population: Treated patients for whom samples were able to be collected
Measure: Geometric Mean (Standard Deviation); unit: ug/L x h
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 17 | 4
ug/L x h | 990 (2.09) | 990 (1.42)

7. Primary Outcome: Elimination Half-life (t 1/2)
Time Frame: Up to 24 hours after dosing
Population: Treated patients for whom PK samples were able to be collected
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 17 | 4
hours | 1.5 (1.3) | 1.5 (1.3)

8. Secondary Outcome: Fludeoxyglucose F18-Positron Emission Tomography Computed Tomography Metabolic Complete Response (mCR) Rate
Description: The mCR rate at recommended phase 2 dose, defined as a metabolic complete response on PET/CT will be defined as greater than -66% reduction in tumor FDG uptake at sites of abnormal tumor FDG uptake noted on pre-treatment FDG-PET study (considering normal cardiac or liver blood pool).
Time Frame: At 3 months post-treatment
Population: Patients who received at least 3 weeks of therapy (cisplatin + triapine), and had their disease re-evaluated with a 3-month post treatment 18F-FDG-PET/CT
Measure: Number (95% Confidence Interval); unit: percentage response-evaluable patients
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 13 | 3
percentage response-evaluable patients | 62 [30 to 86] | 100 [32 to 100]

9. Secondary Outcome: Clinical Overall Response Rate
Description: Clinical response at the recommended phase 2 dose per RECIST v1.1 Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 3 months post-treatment
Population: Patients who received at least 3 weeks of therapy (cisplatin + triapine) and have had their disease re-evaluated (with a 3 month post treatment PET-CT) will be considered evaluable for response. (Note: Patients who exhibit objective disease progression prior to the end of cycle 1 will also be considered evaluable.)
Measure: Number (95% Confidence Interval); unit: percentage response evaluable patient
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 13 | 3
percentage response evaluable patient
  Complete Response | 62 [30 to 86] | 100 [32 to 100]
  Partial Response | 15 [3 to 50] | 0 [0 to 68]
  Stable Disease | 15 [3 to 50] | 0 [0 to 68]
  Progressive Disease | 8 [1 to 42] | 0 [0 to 68]

10. Secondary Outcome: Progression Free Survival (PFS)
Description: Median number of months that patients survive without disease progression from end of treatment. Per RECIST v1.1, Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 4 years and 2 months from start of treatment
Population: Treated patients evaluable for clinical response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 13 | 3
months | NA [NA to NA] — Median not reach due to too few patients experiencing progression | NA [NA to NA] — Median not reach due to too few patients experiencing progression

11. Secondary Outcome: Overall Survival (OS)
Description: Median number of months that patients remain alive after end of treatment.
Time Frame: Up to 4 years and 2 months from start of treatment
Population: Zero treated patients experienced the event of death.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
Number analyzed (Participants) | 17 | 4
months | NA [NA to NA] — not enough events to reach a median | NA [NA to NA] — not enough events to reach a median

ADVERSE EVENTS:
Time Frame: Up to 3 months post-treatment for Adverse Events Up to 4 years and 2 months for All-Cause Mortality
Description: Toxicity evaluated using the NCI CTCAE version 4.0 (version 5.0 beginning April 1, 2018).
Arm/Group | Triapine (100mg) + Chemoradiation) | Triapine (150mg) + Chemoradiation)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/4
Serious Adverse Events (participants affected / at risk) | 8/17 | 2/4
Other Adverse Events (participants affected / at risk) | 17/17 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triapine (100mg) + Chemoradiation) (N=17) | Triapine (150mg) + Chemoradiation) (N=4)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Decreased platelets (Blood and lymphatic system disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Methemoglobinemia (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triapine (100mg) + Chemoradiation) (N=17) | Triapine (150mg) + Chemoradiation) (N=4)
Anemia (Blood and lymphatic system disorders) | 16 | 3
Blood bicarbonate decreased (Blood and lymphatic system disorders) | 1 | 0
Decreased platelets (Blood and lymphatic system disorders) | 13 | 3
Luekocytosis (Blood and lymphatic system disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 2
Sinus bradycardia (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 5 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 6 | 2
Blurred vision (Eye disorders) | 1 | 0
Flashing lights (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Bloating (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhea (Gastrointestinal disorders) | 16 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 15 | 4
Rectal pain (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 3
Chills (General disorders) | 3 | 0
Edema (General disorders) | 4 | 0
Fatigue (General disorders) | 13 | 4
Fever (General disorders) | 2 | 1
Infusion related reaction (General disorders) | 2 | 0
Irritability (General disorders) | 0 | 1
Light headedness (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pelvic infection (Infections and infestations) | 1 | 0
Shingles (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Fogginess (Investigations) | 1 | 1
Increase LDH (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 15 | 4
Methemoglobinemia (Investigations) | 10 | 3
Neutrophil count decreased (Investigations) | 13 | 3
Total protein decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 3 | 1
White blood cell decreased (Investigations) | 14 | 3
Anorexia (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 2
Hypokalemia (Metabolism and nutrition disorders) | 8 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 11 | 3
Hyponatremia (Metabolism and nutrition disorders) | 12 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 1
Restlessness (Psychiatric disorders) | 2 | 0
Bladder pain (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 8 | 2
Hematuria (Renal and urinary disorders) | 6 | 2
Proteinuria (Renal and urinary disorders) | 3 | 0
Urinary frequency (Renal and urinary disorders) | 4 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary pressure (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 2 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 4 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Vaginal bleeding (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 4 | 0
Cold-like symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Perianal sores (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Scrape on knee (Skin and subcutaneous tissue disorders) | 1 | 0
Skin patches (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 1
Hot flashes (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 9 | 1
Hypotension (Vascular disorders) | 1 | 1
Small knots in vein of R leg (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT02595879/Prot_SAP_000.pdf